CLINICAL TRIAL: NCT05461287
Title: An Open-label, Phase 1 Study of QLS31904 as Monotherapy to Assess the Safety, Tolerability and PK in Patients With Advanced Solid Tumors
Brief Title: Safety, Tolerability and Pharmacokinetics Study of QLS31904 in Patients With Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QLS31904-101
Record Dates: First submitted 2022-07-13; First posted 2022-07-18 (Actual); Last update posted 2022-11-10 (Actual); Status verified 2022-11

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- QLS31904 (Experimental): Qls31904 is a bi-specific recombinant protein construct containing 2 humanized antibody derived binding domains.
  Interventions: Drug: QLS31904

INTERVENTIONS:
Drug: QLS31904 — QLS31904 ONLY

SUMMARY:
This is an open label, phase 1 clinical study to evaluate the safety, tolerability, dose limiting toxicities (DLTs), maximum tolerated dose (MTD) or maximum administered dose (MAD) and recommended phase 2 dose (RP2D) of QLS31904 q2w/q3w intravenous use in patients with advanced solid tumors. Additional objectives are to characterise pharmacokinetics and pharmacodynamics, and to evaluate efficacy signals. This study is consisted of phase Ia (Dose Escalation) and phase Ib (Dose Expansion). Phase Ib will further explore QLS31904 in selected patients populations based on data from phase Ia. The Phase Ib objectives, endpoints and design will be specified in a study protocol amendment after availability of phase Ia results.

ELIGIBILITY:
Inclusion Criteria:

1. Understanding and voluntarily signing the informed consent form;
2. Male or female, age≥18 years;
3. Patients with histologically or cytologically confirmed advanced solid tumors including small cell lung cancer, small cell cancers in other organs or neuroendocrine carcinoma who have progression after on theor intolerance to standard of care, or have no effective standard therapeutic regimen;
4. Tumours must be confirmed expression of DLL3.
5. Presence of at least one measurable lesion meeting the requirements in RECIST v1.1 evaluation criteria;
6. ECOG PS score: 0~1;
7. Patients with life expectancy ≥3 months;
8. Adequate organ function as defined in protocol. Futher inclusion criteria apply.

Exclusion Criteria:

1. Having received the treatment targeting CD3 or DLL3 previously;
2. Receiving any systematic antitumor therapy or other investigational product within 4 weeks prior to the first dose of QLS31904;
3. Receiving radiotherapy within 2 weeks prior to the first dose of QLS31904;
4. For the dose-escalation, participants who experienced severe immune-mediated AEs while on treatment with Immune checkpoint inhibitors (e.g., anti PD-L1, anti PD-1, anti CTLA-4) ;
5. Symptomatic central nervous system (CNS) metastasis.
6. History of concurrent serious cerebro- and cardiovascular diseases including but not limited to: unstable angina pectoris, myocardial infarction, cerebrovascular accident or transient ischemic attack within 6 months prior to the first doses, poorly controlled hypertension or arrhythmia, or any other arterial thrombosis or embolic event;
7. History of concurrent gastrointestinal diseases including but not limited to: gastrointestinal bleeding or perforation, acute pancreatitis;
8. History of concurrent lung damage including but not limited to: interstitial lung disease, other diseases requiring oxygen inhalation.
9. Presence of active pneumonia or history of noninfectious pneumonia;
10. Active infection requiring systematic treatment/antibiotics or intravenous use of systemic anti-infection therapy with one week prior to the first dose or use for more than 7 days;
11. Known positive for human immunodeficiency virus (HIV); Having evidence on infection of hepatitis C virus (HCV) or syphilis; Hepatitis B virus (HBV) infected individuals with positive HBsAg and HBV DNA copy >1000 IU/ml or 200 cps/mL; Following treatment according to guidelines, previously HBV infected individuals in screening period can be enrolled only;
12. Presence of active or suspicious autoimmune disease.
13. Previous allogeneic bone marrow transplantation or solid organ transplantation;
14. Major surgery (judged by investigators) or in the recovery period of the surgery within 4 weeks before the first dose of QLS31904.
15. Vaccination of live attenuated vaccine within 4 weeks prior to the first dose of QLS31904;
16. Having other malignant tumor other than the disease investigated within 2 years prior to the ICF;
17. Known allergy to any component of QLS31904;
18. Any other disease or condition of clinical significance that can affect the compliance with the protocol (e.g., history of psychosis or drug abuse), affect the signature of the informed consent form (e.g., drug addiction and drug abuse);
19. Any condition is unsuitable to be involved in this clinical trial, as considered by investigators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 290 (Estimated)
Dates: Start 2022-09-30 (Actual); Primary Completion 2024-09-25 (Estimated); Study Completion 2025-05-25 (Estimated)

PRIMARY OUTCOMES:
DLT | Up to 28 approximately days
  Dose-limiting toxicity (DLT) is defined as any of the specified toxicities evaluated as at least possibly related with the study drug within 28 days after the first dose.
MTD | Up to 24 approximately months
  The maximum tolerated dose (MTD) is defined as the highest dose at which DLT occurs in <1/3 subjects.
  The maximum administrated dose (MAD) is defined as the highest dose of all groups if MTD can not be determined.
RP2D | Up to 24 approximately months
  Recommended dose for phase II trials

SECONDARY OUTCOMES:
Incidence of adverse event (AE) | Up to 24 approximately months
  Incidence of adverse events (AE) assessed according to NCI-CTCAE 5.0 Incidence of adverse events (AE) assessed according to NCI-CTCAE 5.0
Severity of adverse event (AE) | Up to 24 approximately months
  Severity of adverse events (AE) assessed according to NCI-CTCAE 5.0
Incidence of serious adverse event (SAE) | Up to 24 approximately months
  Incidence of serious adverse event (SAE) assessed according to NCI-CTCAE 5.0
Severity of serious adverse event (SAE) | Up to 24 approximately months
  Severity of serious adverse events (AE) assessed according to NCI-CTCAE 5.0
Incidence of immune related adverse event (irAE) | Up to 24 approximately months
  Incidence of immune related adverse event (irAE) assessed according to NCI-CTCAE 5.0
Incidence of clinically significant laboratory examination and abnormal changes in other examinations | Up to 24 approximately months
  Incidence of clinically significant laboratory examination and abnormal changes in other examinations assessed according to NCI-CTCAE 5.0
peak concentration (Cmax) | Up to 24 approximately months
  Pharmacokinetic (PK) profile: drug concentration in individual subject at different time points after administration; pharmacokinetic parameters peak concentration (Cmax);
time to peak (Tmax) | Up to 24 approximately months
  Pharmacokinetic (PK) profile: drug concentration in individual subject at different time points after administration; pharmacokinetic parameters time to peak (Tmax);
trough concentration (Ctrough) | Up to 24 approximately months
  Pharmacokinetic (PK) profile: drug concentration in individual subject at different time points after administration; pharmacokinetic parameters trough concentration (Ctrough)
area under the plasma drug concentration-time curve (AUC0-t ) | Up to 24 approximately months
  Pharmacokinetic (PK) profile: drug concentration in individual subject at different time points after administration; pharmacokinetic parameters area under the plasma drug concentration-time curve (AUC0-t )
area under the plasma drug concentration-time curve (AUC0-inf) | Up to 24 approximately months
  Pharmacokinetic (PK) profile: drug concentration in individual subject at different time points after administration; pharmacokinetic parameters area under the plasma drug concentration-time curve (AUC0-inf);
volume of distribution (Vss) | Up to 24 approximately months
  Pharmacokinetic (PK) profile: drug concentration in individual subject at different time points after administration; pharmacokinetic parameters volume of distribution (Vss)
elimination half-life (t1/2) | Up to 24 approximately months
  Pharmacokinetic (PK) profile: drug concentration in individual subject at different time points after administration; pharmacokinetic parameters elimination half-life (t1/2)
clearance rate (CL) | Up to 24 approximately months
  Pharmacokinetic (PK) profile: drug concentration in individual subject at different time points after administration; pharmacokinetic parameters clearance rate (CL);
mean retention time (MRT) | Up to 24 approximately months
  Pharmacokinetic (PK) profile: drug concentration in individual subject at different time points after administration; pharmacokinetic parameters mean retention time (MRT)
ORR | Up to 24 approximately months
  The efficacy evaluated by the investigator in accordance with RECIST 1.1 criteria, including objective response rate (ORR).
DOR | Up to 24 approximately months
  The efficacy evaluated by the investigator in accordance with RECIST 1.1 criteria24, including duration of response (DOR);
DCR | Up to 24 approximately months
  The efficacy evaluated by the investigator in accordance with RECIST 1.1 criteria24, including disease control rate (DCR);
PFS/PFS6 | Up to 24 approximately months
  The efficacy evaluated by the investigator in accordance with RECIST 1.1 criteria24, including progression-free survival (PFS) and percents of progression-free survival more than six months;
OS | Up to 24 approximately months
  The efficacy evaluated by the investigator in accordance with RECIST 1.1 criteria24, including overall survival (OS);
ADA | Up to 24 approximately months
  incidence of anti-drug body (ADA)
Nab | Up to 24 approximately months
  concentration of neutralizing antibody (Nab);

OTHER OUTCOMES:
DLL3 expression in tumor tissue | Up to 24 approximately months
  To explore the correlation between DLL3 expression in tumor tissue and the efficacy
Objective response based on iRECIST criteria in patients with measurable disease | Up to 24 approximately months
  Objective response based on immune Response Evaluation Criteria in Solid Tumors (iRECIST) criteria in patients with measurable disease

CONTACTS AND LOCATIONS:
Locations (1):
- Jilin Cancer Hospital, Changchun, Jilin, China